CLINICAL TRIAL: NCT00987441
Title: Epidural Analgesia for Labor Pain and Infant Neurobehavior
Brief Title: Epidural Labor Analgesia and Infant Neurobehavior
Acronym: ELAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NJMU-0933MZ; NMUK2191
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Labor Pain
Keywords: Neurobehavior; Epidural analgesia; Local anesthetic; Opioid
MeSH Terms: conditions — Labor Pain | interventions — Ropivacaine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Local anesthetic plus opioid 1 (Active Comparator): Local anesthetic (ropivacaine 0.125%) plus first opioid dose (sufentanil 0.3 microgram/ml) delivered peridural space
  Interventions: Drug: Ropivacaine and sufentanil
- Local anesthetic plus opioid 2 (Active Comparator): Local anesthetic (ropivacaine 0.125%) plus second opioid dose (sufentanil 0.4 microgram/ml) delivered peridural space
  Interventions: Drug: Ropivacaine and sufentanil
- Local anesthetic plus opioid 3 (Active Comparator): Local anesthetic (ropivacaine 0.125%) plus third opioid dose (sufentanil 0.5 microgram/ml) delivered peridural space
  Interventions: Drug: Ropivacaine and sufentanil
- Local anesthetic 1 plus opioid (Active Comparator): First local anesthetic dose (ropivacaine 0.0625%) plus opioid (sufentanil 0.4 microgram/ml) delivered peridural space
  Interventions: Drug: Ropivacaine and sufentanil
- Local anesthetic 2 plus opioid (Active Comparator): Second local anesthetic dose (ropivacaine 0.1875%) plus opioid (sufentanil 0.4 microgram/ml) delivered peridural space
  Interventions: Drug: Ropivacaine and sufentanil
- Local anesthetic 3 plus opioid (Active Comparator): Third local anesthetic dose (ropivacaine 0.25%) plus opioid (sufentanil 0.4 microgram/ml) delivered peridural space
  Interventions: Drug: Ropivacaine and sufentanil

INTERVENTIONS:
Drug: Ropivacaine and sufentanil — Ropivacaine 0.125% plus sufentanil 0.3 microgram
  Other Names: Naropin; Sufenil
  Arms: Local anesthetic plus opioid 1
Drug: Ropivacaine and sufentanil — Ropivacaine 0.125% plus sufentanil 0.4 microgram
  Other Names: Naropin; Sufenil
  Arms: Local anesthetic plus opioid 2
Drug: Ropivacaine and sufentanil — Ropivacaine 0.125% plus sufentanil 0.5 microgram
  Other Names: Naropin; Sufenil
  Arms: Local anesthetic plus opioid 3
Drug: Ropivacaine and sufentanil — Ropivacaine 0.0625% plus sufentanil 0.4 microgram
  Other Names: Naropin; Sufenil
  Arms: Local anesthetic 1 plus opioid
Drug: Ropivacaine and sufentanil — Ropivacaine 0.1875% plus sufentanil 0.4 microgram
  Other Names: Naropin; Sufenil
  Arms: Local anesthetic 2 plus opioid
Drug: Ropivacaine and sufentanil — Ropivacaine 0.25% plus sufentanil 0.4 microgram
  Other Names: Naropin; Sufenil
  Arms: Local anesthetic 3 plus opioid

SUMMARY:
Infant neurobehavior alteration is predictor of later intelligence development. Many factors would influence or are associated with infant neurobehavior, of which exist or appear during perinatal period. Neuraxial, especially epidural, analgesia to date is the most effective method in relieving labor pain. Although previous studies showed that opioid used in epidural analgesia for labor pain can affect newborn neurobehavior negatively in a dose-escalation associated manner, whether epidural analgesia itself would produce unpredictable effect on newborn neurobehavior is still unknown. Hereby the investigators designed this trial to investigate the hypothesis that epidural analgesia for labor pain control itself would not produce negative effect on infant neurobehavior.

ELIGIBILITY:
Inclusion Criteria:

* >18years and <45years
* Spontaneous labor
* Analgesia request

Exclusion Criteria:

* Allergy to opioids, a history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records
* Participants younger than 18 years or older than 45 years
* Those who were not willing to or could not finish the whole study at any time
* Using or used in the past 14 days of the monoamine oxidase inhibitors
* Alcohol addictive or narcotic dependent patients were excluded for their influence on the analgesic efficacy of the epidural analgesics
* Subjects with a nonvertex presentation or scheduled induction of labor

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | Immediate after birth (0 min)

SECONDARY OUTCOMES:
Apgar scoring | One min and 5min after birth.
Umbilical-cord gases analysis | At the time baby was born (0min)
Neonatal sepsis evaluation | One hour after the baby was born
Neonatal antibiotic treatment | One hour after the baby was born
Incidence of maternal side effects | Analgesia initiation (0min) to successful vaginal delivery (this time encountered alteration with different women)
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 10min after birth
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 1h after birth
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 8h after birth
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 1d after birth
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 1wk after birth

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- The Affiliated Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China